CLINICAL TRIAL: NCT06495294
Title: SWiFT Canada (Study of Whole Blood in Frontline Trauma): A Pilot Randomized Controlled Trial Assessing Prehospital Whole Blood Versus Component Therapy in Traumatic Hemorrhage
Brief Title: SWiFT Canada (Study of Whole Blood in Frontline Trauma)
Acronym: SWiFTCanada
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Veteran Affairs Canada (Unknown); Ornge (Unknown); Canadian Blood Services (Other); Sunnybrook Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other); London Health Sciences Centre (Other); Kingston Health Sciences Centre (Other); Health Sciences North (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-4921
Record Dates: First submitted 2024-06-05; First posted 2024-07-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Trauma
Keywords: prehospital; major hemorrhage; transfusion; emergency medicine
MeSH Terms: conditions — Wounds and Injuries | interventions — Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: A multicentre, pragmatic, randomized controlled, open-label, parallel group two arm trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Blood (WB) (Experimental): The use of Whole Blood (WB), leukocytes reduced is indicated for treatment of patients with clinically significant bleeding and have low anti-A and anti-B titres.
  Patients will be administered up to 2 units of whole blood administered via either intravenous (IV) or intraosseous (IO) route, according to standard practice at Ornge AAS.
  Interventions: Biological: Whole Blood
- Red Blood Cells and Plasma (Active Comparator): The control arm will consist of 2 units of RBC and 2 units of plasma (dependent on the standard practice of the Ornge AAS).
  RBC and plasma may be administered via either the intravenous (IV) or intraosseous (IO) route, according to standard clinical practice at Ornge AAS.
  Interventions: Biological: RBC + plasma

INTERVENTIONS:
Biological: Whole Blood — 2 units of whole blood administered by Ornge AAS
  Arms: Whole Blood (WB)
Biological: RBC + plasma — 2 units of RBC + 2 units of plasma administered by Ornge AAS
  Arms: Red Blood Cells and Plasma

SUMMARY:
Traumatic injuries affect people of all ages, races, and socioeconomic backgrounds. The Global Burden of Disease study showed that globally in 2019, there were more than 4.4 million deaths due to injury. Furthermore, unintentional injuries are the leading cause of death for people aged 5-29 years worldwide. Uncontrolled bleeding accounts for a significant proportion of these deaths, with approximately 20% occurring in the first 24 hours and 40% occurring within the first 30 days.

Blood transfusion is a life-saving treatment in the management of bleeding patients until bleeding is controlled in hospital, typically delivered through different blood components (red blood cells, plasma and platelets). These components are derived from a whole blood donation and are stored in separate bags (units). There are challenges in carrying separate blood products, such as additional weight in kit bags, and transfusing multiple blood products at the scene can delay transport to hospital.

In Ontario, Ornge Air Ambulance carries red blood cells and plasma to transfuse prehospital. However, a prehospital transfusion strategy has not been established and practice varies across the Canadian setting, and more broadly across the world.

This trial aims to investigate if carrying and transfusing two units of whole blood instead of four units (two red blood cells and two plasma) is feasible and leads to better outcomes for patients.

DETAILED DESCRIPTION:
Early blood transfusion improves survival in patients with life-threatening bleeding, but the optimal transfusion strategy in the prehospital setting has yet to be established. Although there is some evidence of benefit with the use of Whole Blood (WB), there have been no RCTs exploring the clinical effectiveness of prehospital administration of WB versus component therapy for bleeding trauma patients in the Canadian setting. The lack of high-quality clinical evidence is recognized in the recent NAC recommendations for the use of WB in Canada.

In collaboration with the SWiFT UK team, the SWiFT Canada study will follow the SWiFT UK protocol but as adopted for the Canadian context. This may allow for future comparisons on effectiveness of the two systems and pilot the ability for two countries with different prehospital systems to be able to follow a similar study protocol for future international RCTs.

Lastly, we have confirmed the support from CBS for the manufacturing and distribution of WB for the duration of the SWiFT Canada trial. Therefore, it is essential for patients, healthcare professionals and blood services that the clinical effectiveness of prehospital WB transfusion is evaluated in a trial before its widespread implementation across CBS in Canada. A national program of WB production would necessitate significant changes in the current manufacturing processes for blood services, in order to provide appropriate support for hospitals. WB production could potentially affect the supply of blood components required to treat other patients, as a unit of WB cannot be used to manufacture other components. However, it could also be argued that early transfusion of WB may reduce the need for further blood component transfusion when patients arrive at hospital, due to earlier control of bleeding. Following the proposed objectives of this pilot RCT would enable us to evaluate all these uncertainties and assist in the planning of a future larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has suffered a traumatic injury
* Attended by a participating Ornge AAS clinical team
* Requires prehospital blood transfusion to treat major traumatic hemorrhage

Exclusion Criteria:

* Pediatric (age <16 or transported to pediatric trauma centre [if age unknown])
* No intravenous or intraosseous access (should be assessed prior to opening box)
* Knowledge that patient will object to being given blood transfusion for any reasons
* Blood already administered on-scene, prior to arrival of the participating Ornge AAS

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients enrolled in the study that receive a prehospital transfusion and had full study data collected | through study completion, up to 90 days
  Feasibility target: >90% patients enrolled were able to link prehospital to in-hospital records and >90% complete data obtained
Number of patients that completed transfusion of at least 1 unit of assigned blood products prior to arrival to receiving lead trauma hospital | Enrolment to day 1 after enrolment
  Feasibility target: at least 1 unit of blood [WB, RBC, or plasma] transfused prior to arrival >90% of the time
Number of patients that completed transfusion of all assigned blood products at the receiving lead trauma hospital | Enrolment to day 1 after enrolment
  Feasibility target: >90% if not already done prior to arrival of hospital
Number of patients screened for the study by not randomized due to lack of group O negative WB availability. | through study completion, an average of 1 year
To describe the distribution, redistribution and wastage of WB units produced for the study | through study completion, an average of 1 year
  Feasibility target: <10% wastage of WB units produced for the study

SECONDARY OUTCOMES:
Death or Massive Transfusion at 24hrs | through study completion, up to 90 days
  To determine the impact of prehospital administration of WB on the proportion of participants who experience death or massive transfusion at 24 hours, compared to the current standard of care (component blood therapy).
Mortality - 90 days | through study completion, up to 90 days
  To determine the impact on mortality up to 90 days.
Mortality - 30 days | through study completion, up to 90 days
  To determine the impact on morbidity up to 30 days.
Organ Failure Free Days | through study completion, up to 90 days
  To determine the impact of organ failure free days (hospital resource use) up to discharge
Critical Care Days | through study completion, up to 90 days
  To determine the impact of time spent in critical care (hospital resource use) up to discharge
Total in-patient stay | through study completion, up to 90 days
  To determine the impact on total in-patient stay (hospital resource use) up to discharge
Blood components received | through study completion, up to 90 days
  To determine the impact on blood components received (hospital resource use) up to discharge
Hemostatic agents received | through study completion, up to 90 days
  To determine the impact additional hemostatic agents received (hospital resource use) up to discharge
treatment-emergent adverse events | through study completion, up to 90 days
  To assess the safety and tolerability of prehospital transfusion by the incidence of treatment-emergent transfusion adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Brodie Nolan, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- Ornge Air Ambulance, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publish study protocol, including statiscal analysis plan, informed consent process
Supporting Information: Study Protocol
Time Frame: Starting in September 2024, protocol will be available.
Access Criteria: Please contact the trial leadership at swift@unityhealth.to
URL: https://first60.ca/current-studies/swift/

REFERENCES:
- [Derived] Lin Y, Peddle M, Callum J, Beckett A, da Luz LT, Drennan I, Pavenski K, Mack J, McGowan M, Ahghari M, Smith J, Green L, Keown-Stoneman CDG, Nolan B; SWiFT Canada Investigators. Study protocol for a pilot randomised controlled trial assessing prehospital whole blood versus component therapy in traumatic haemorrhage: SWiFT Canada (study of whole blood in frontline trauma). BMJ Open. 2025 Dec 31;15(12):e108570. doi: 10.1136/bmjopen-2025-108570. PMID 41475814
- See also: SWiFT Canada Study Site — https://first60.ca/current-studies/swift/